CLINICAL TRIAL: NCT00739895
Title: Left Ventricular Dilatation in Athletes With Common Colds; a Cardio-vascular MRI Study
Brief Title: Assessment of Cardiac Involvement of Common Cold in High Performing Athletes by Cardiac Magnetic Resonance Imaging (MRI)
Status: Terminated | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Oliver Strohm, adunct Research Associate Professor, University of Calgary
Other Study IDs: Athletes_001
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Ventricular Function, Left
Keywords: athletes
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Athletes: high performing athletes
  Interventions: Procedure: Cardiac magnetic Resonance study; Procedure: Blood testing

INTERVENTIONS:
Procedure: Cardiac magnetic Resonance study — follow-up studies
Procedure: Blood testing — Blood sample tested for myocardial biomarkers

SUMMARY:
Cardiovascular magnetic resonance (CMR) imaging will be used to assess the impact of common colds and physical training in high-performing athletes. Healthy individuals from the general public will serve as a comparison group. CMR has previously been shown to accurately assess cardiac function, edema, inflammation, and injury.

Athletes competing at National level and Developmental Canadian teams will be prospectively recruited. All participants will have CMR scans at low and high intensity training. Participants will be re-scanned immediately after clinical evidence of a common cold, as determined by respiratory and flu-like symptoms. After 4 weeks, a follow-up CMR scan will be performed. On the day of each CMR scan, electrocardiograms and blood samples will be drawn from each participant. Blood samples will provide markers of systemic inflammation, such as leukocyte counts. At each CMR scan, athletes will be asked to describe there recent history of physical exertion in questionnaires, which will reflect the degree of physical exertion performed.

DETAILED DESCRIPTION:
Cardiovascular magnetic resonance (CMR) imaging will be used to assess the impact of a common colds and physical training in high-performing athletes. Healthy individuals from the general public will serve as a comparison group. CMR has previously been shown to accurately assess cardiac function, edema, inflammation, and injury.

Athletes competing at National level and Developmental Canadian teams will be prospectively recruited. All participants will have CMR scans at low and high intensity training. Participants will be re-scanned immediately after clinical evidence of a common cold, as determined by respiratory and flu-like symptoms. After 4 weeks, a follow-up CMR scan will be performed. On the day of each CMR scan, electrocardiograms and blood samples will be drawn from each participant. Blood samples will provide markers of systemic inflammation, such as leukocyte counts. At each CMR scan, athletes will be asked to describe there recent history of physical exertion in questionnaires, which will reflect the degree of physical exertion performed.

Image analysis: CMR parameters that serve as surrogate markers for myocardial inflammation will be assessed. Specifically, they include STIR (edema), early enhancement (inflammation), and late enhancement (fibrosis). The presence of 2 of these parameters will indicate the presence of myocardial inflammation. Qualitative and quantitative analysis will be performed on images obtained from CMR scans, and will be assessed offline using CMR42 (Circle International, Calgary) software. Standard methods of assessing edema, inflammation, and fibrosis will be implemented. Standard left ventricular function volume analysis techniques will be implemented to assess left ventricular dilatation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent;
* feverish feeling with last 72 hours;
* active participation in competitive sports;
* history of recent viral exposure or flu-like symptoms.

Exclusion Criteria:

* CMR Contraindications,
* chronic diseases affecting the heart,
* use of immuno-active drugs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: high performance athletes, during acute viremia and at variable training intensities. Healthy individuals from the general public will serve as a reference group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Left-ventricular systolic dysfunction, as defined by increased left ventricular end-diastolic volume | 12 months

SECONDARY OUTCOMES:
Myocardial edema, fibrosis, inflammation, volumetry | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias G Friedrich, MD, FESC, Principal Investigator — University of Calgary
Locations (1):
- Stephenson CMR Centre at Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada